CLINICAL TRIAL: NCT05795673
Title: Peer-supporting for Teenagers With Cystic Fibrosis in a Process of Transition of Care From Paediatric to Adult Services : a Mixed-method Pilot Study to Assess the Feasibility of the Peer-support Intervention
Brief Title: Peer-supporting for Teenagers With Cystic Fibrosis in the Transition of Care From Paediatric to Adult Services
Acronym: MUKADO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 69HCL21_1096
Record Dates: First submitted 2023-02-02; First posted 2023-04-03 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Peer helping; Transition
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Intervention Model Description: Prospective quasi-experimental before-and-after multicenter study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Peer support (Other): Intervention of mentor to provide peer support
  Interventions: Other: Peer support program (intervention phase)
- Group Control (No Intervention): Usual practices of accompaniment of the pediatric-adult transition

INTERVENTIONS:
Other: Peer support program (intervention phase) — Implementation and Evaluation:
  Intervention of mentor to provide peer support targeting psychosocial skills, coping and quality of life of adolescents with cystic fibrosis during the pediatric-adult transition The evaluation of the feasibility of the peer support program consists of assessing the effectiveness of its implementation in terms of its effect on the target audience, its acceptability to participants, and its implementation.
  The mentor and the mentee will be in contact once a month for a minimum of 3 months and a maximum of 6 months by telephone.
  The mentor will know the themes that the teenager would like to address in the context of peer support.
  The mentee will complete the various questionnaires provided in the protocol to answer the primary and secondary endpoints.
  Arms: Group Peer support

SUMMARY:
In patients with cystic fibrosis, a deterioration in lung function around age 18, the age of transfer from pediatrics to adult care services, has been observed. Transfer is only one step in a transition process from pediatric to adult care taking place from age 12 to 24. Adolescence is a period of identity construction during which the disease alters self-image and self-esteem, and a period of empowerment in the management of the disease involving a re-appropriation of it. During this period, coping strategies and psychosocial skills are important to face all the issues that the adolescent encounters. Interventions for youth with chronic illnesses rarely incorporate this dimension. Peer support or peer-mentoring is one avenue for developing these coping skills. Peer support encompasses mutual support between people who are coping or have coped with similar challenging life experiences. Individuals with similar experiences would represent more credible role models to stimulate positive change in their peers. The function of peer support are to provide emotional, experiential, informational support.The effect of peer support improves social integration, coping skills, sense of self-efficacy of the peers being helped. Promotion of healthy youth behaviors by youth is the most widely evaluated youth engagement strategy in the community health sector. Peer-assisted devices have been tested to improve medication adherence and health status with youth with juvenile arthritis, asthma, and liver transplant recipients. By sharing their experience of a successful transition, young adults with cystic fibrosis may be able to help their adolescent peers better understand this transition. Our hypothesis is that implementing peer support with adolescents with cystic fibrosis improves their sense of self-efficacy, a dimension of coping skills.To our knowledge, there are no research studies on peer support in cystic fibrosis in France or abroad. Patients are recognized as partners capable of sharing their experiential knowledge with patients with a similar disease.

But this raises questions about the recruitment, supervision, preparation for peer-help and the role of these patients; about the effects of their involvement for themselves (valorization, anxiety) and for their peers (re-assurance, feeling of personal effectiveness). This justifies conducting an exploratory study to assess the feasibility of a peer-support intervention for youth with cystic fibrosis.

ELIGIBILITY:
Concerning the patient /mentee:

Inclusion Criteria:

* patient affected by cystic fibrosis
* patient able to understand and read French
* patient from 15 to 19 years , in a process of transition on paediatric care to adult care
* with a follow-up on a paediatric Cystic Fibrosis Centers Competences (CRCM)
* did not participate in the Phase 1 co-construction workgroup
* affiliated to the social security system
* having agreed to participate and signed the consent for an adult patient, or legal guardian having agreed to participate and signed the consent for a minor patient

Exclusion Criteria:

* patient with transplant
* patient with cystic fibrosis transmembrane regulator-related disorders (CFTR RD) or Screen Positive Inconclusive Diagnosis (SPID) Cystic Fibrosis
* patient with a curator, tutor or under the protection of a conservator
* pregnant or breastfeeding patient

Concerning the mentor/peer-supporter (post period):

Inclusion Criteria * :

* affected cystic fibrosis
* able to understand and read French
* young adult, 19 to 24 years old
* with a follow-up on the adult CRCM (transition completed)
* affiliated to the social security system
* have agreed to participate and signed the consent form
* did not participate in the Phase 1 co-construction workgroup

Exclusion Criteria * :

* patient with transplant
* patient with CFTR RD or SPID Cystic Fibrosis
* patient with a curator, tutor or under the protection of a conservator
* pregnant or breastfeeding patient

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 88 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Quality of life of adolescents in transition, measured by the French version of the Cystic Fibrosis Questionnaire - Revised (CFQ-R) at 6 months | Baseline ; at 6 months
  Change in Quality of life of adolescents in transition, measured by the French version of the Cystic Fibrosis Questionnaire - Revised (CFQ-R) at 6 months. The CFQ-R includes 34 cystic fibrosis-specific quality of life items, scored on a 4-modality scale, and exploring 9 dimensions including perceived health, burden of treatment, self-image (and body image in particular), emotional state, and social interaction that are particularly impacted by the transition period. The responses allow us to establish a score on a scale of 0 to 100, the higher the score the better the quality of life.
Change from baseline Quality of life of adolescents in transition, measured by the French version of the Cystic Fibrosis Questionnaire - Revised (CFQ-R) at 3 months | Baseline ; at 3 months
  Change in Quality of life of adolescents in transition, measured by the French version of the Cystic Fibrosis Questionnaire - Revised (CFQ-R) at 3 months. The CFQ-R includes 34 cystic fibrosis-specific quality of life items, scored on a 4-modality scale, and exploring 9 dimensions including perceived health, burden of treatment, self-image (and body image in particular), emotional state, and social interaction that are particularly impacted by the transition period. The responses allow us to establish a score on a scale of 0 to 100, the higher the score the better the quality of life.

SECONDARY OUTCOMES:
Effect of peer support model during pediatric-adult transition, assessed in adolescents (comparison between sponsored adolescents and non-sponsored adolescents) on their sense of self-efficacy | Measurement at inclusion, 3 months and 6 months
  Adolescents' sense of self-efficacy (Phase 2 primary endpoint), measured by the French version of the generic 10-item General Self-Efficacy Scale (GSE) rated on a 4-modality scale (not at all true, barely true, moderately true, totally true).
Effect of peer support model during pediatric-adult transition, assessed in adolescents (comparison between sponsored adolescents, included in post period, and non-sponsored adolescents, included in pre period) on management and therapeutic adherence | Measurement at inclusion, 3 months and 6 months
  Management and therapeutic adherence, measured by a cystic fibrosis-specific adherence self-assessment questionnaire and focusing on the patient's perceived adherence to the respiratory (physical therapy and therapeutics), digestive and nutritional components of cystic fibrosis management. This Cystic Fibrosis Compliance questionnaire will be used in its French version. Indeed, it has already been translated according to a standard translation-re translation procedure by the same research study in a previous study (N° 2019-A01029-48, favorable opinion of the Ethic committee West IV - Nantes on 10/09/2019). This previous study is still in progress and will be published at the end of the study.
Effect of peer support model during the pediatric-adult transition, assessed in adolescents (comparison between sponsored adolescents, included in the post period, and non-sponsored adolescents, included in the pre period) on sense of social integration. | Measurement at inclusion, 3 months and 6 months
  Sense of social integration, measured by the 5 items of the "social integration and support" dimension of the validated French version of the Health Education Impact Questionnaire (heiQ).
  The items are: 22) If I need help, I have people I can count on; 28) I have enough friends to help me cope with my health problems;31) When I feel sick, my family and the people who take care of me understand what I am going through;35) In general, I feel that my friends and family look after me well;37) I have enough opportunities to talk about my health problems with people who understand me. Responses are rated on a 4-way agreement scale (strongly disagree, disagree, agree, strongly agree).
Fidelity of peer-assistance process in relation to what was planned (criteria collected in the "after" period only). | From inclusion to the end of pair-aidance, up to 8 months
  Fidelity of the peer-assistance process in relation to what was planned (criteria collected in the "after" period only):
  Collection of implementation indicators (grid for collecting the number of contacts between sponsor and sponsored person, the modalities and the themes discussed during the contacts) and qualitative analysis of the content of the exchanges of practices between sponsors during the peer-assistance period.
Experience (Experience, Satisfaction, Acceptability) of peer support among sponsored adolescents, sponsors, parents and accompanying professionals by individual interviews 1 to 2 months after the end of peer support (collected in the "after" period). | From inclusion to the end of pair-aidance, up to 8 months
  Perceived experience/other effects of peer support by the accompanying professionals, and in particular perceived effects of peer support on their clinical practice.
  * Experience/other perceived effects of peer support by sponsored adolescents, sponsors, parents.
  * Acceptability and satisfaction of peer support by the participants (sponsored adolescents, sponsors, parents and accompanying professionals): Satisfaction feedback and identification of factors influencing acceptability (participants' sociodemographic characteristics, patients' clinical characteristics, sponsors' previous experiences of supportive roles, status and experiences of accompanying professionals, characteristics of the CRCM).
  The collection and analysis of these three criteria will be carried out by means of a qualitative study using individual semi-directed interviews (criteria collected in the "after" period only), the content of which will be developed in phase 1.
Feasibility assessed by the number of questionnaires collected | From inclusion to the end of pair-aidance, up to 8 months
  Feasibility will be validate if a minimum of 90 questionnaires is collected
Feasibility assessed by the estimation of recruitment capacity | From inclusion to the end of pair-aidance, up to 8 months
  Recruitment capacity will be validate if a minimum of 30 patients (15 during each period) is included
Feasibility assessed by the number of resources needed to implement the intervention - Number and profile of accompanying professionals involved | From inclusion to the end of pair-aidance, up to 8 months
  Collection of the profesionnel's profile implicated on the study
Feasibility assessed by the number of resources needed to implement the intervention - Number of exchanges and time needed for supervision and training | From inclusion to the end of pair-aidance, up to 8 months
  Tracking of exchange and the necessary time for training
Feasibility assessed by the number of resources needed to implement the intervention - Collection of material resources needed | From inclusion to the end of pair-aidance, up to 8 months
  Peer support constructed during the period 1
Feasibility assessed by the estimation of the potential effect of the intervention on the feeling of self-efficacy measured by the GSE | From inclusion to the end of pair-aidance, up to 8 months
  The generic 10-item GSE rated on a 4-modality scale (not at all true, barely true,moderately true, totally true).
  The total score is calculated by finding the sum of the all items. For the GSE, the total score ranges between 10 and 40, with a higher score indicating more self-efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Quitterie REYNAUD, MD, Principal Investigator — Hospices Civils de Lyon
Locations (4):
- France (4):
  - CRCM Lyon pédiatrie - Hôpital Femme Mère Enfant, Hospices Civils de Lyon, Bron
  - CRCM Grenoble adulte - Hôpital Albert Michallon, Grenoble
  - CRCM Grenoble pédiatrie - Hôpital Albert Michallon, Grenoble
  - CRCM Lyon adulte - Centre Hospitalier Lyon Sud, Hospices Civils de Lyon, Pierre-Bénite